CLINICAL TRIAL: NCT03255161
Title: Oyendo Bien: Reducing Disparities in Access to Hearing Health Care on the U.S.-Mexico Border
Brief Title: Randomized Controlled Trial of a Community Health Worker Program on Hearing Loss (Oyendo Bien)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Arizona (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: UArizona1; R33DC013681 (NIH)
Record Dates: First submitted 2017-08-14; First posted 2017-08-21 (Actual); Last update posted 2019-10-07 (Actual); Status verified 2018-10

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss | interventions — Self-Help Groups

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate communication education and support group (Experimental)
  Interventions: Behavioral: community health worker-audiologist communication education and support group
- Waitlist (No Intervention)

INTERVENTIONS:
Behavioral: community health worker-audiologist communication education and support group — A 5-week educational program on hearing loss, communication strategies, and peer support facilitated by community health workers supervised by an audiologist.
  Arms: Immediate communication education and support group

SUMMARY:
The purpose of this study is to test the effectiveness of a community health worker intervention to expand access to hearing health care among older adults facing health disparities.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age: 50 years
* Audiometrically-confirmed hearing loss
* Availability of a communication partner to attend the program with the participant
* Be Spanish speaking and able to sign written informed consent

Exclusion Criteria:

* Cognitive impairment

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-08-19 (Actual); Primary Completion 2019-01-23 (Actual); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
Mean frequency of communication strategy use as measured at eight weeks post baseline for each of a series of study-specific strategies taught in the intervention | 8 weeks
  Participants rate the frequency of use of each communication strategy on a five-point Likert scale. Communication strategies include such things as discussing hearing loss, talking face-to-face, and speaking slowly and clearly.

SECONDARY OUTCOMES:
Mean number of hearing health actions taken and number of people who took each hearing health action at eight weeks post baseline | 8 weeks
  Questionnaire includes 7 possible actions for managing hearing health or accessing hearing health care services (discussed with family, discussed with doctor, discussed with specialist, had a hearing test, used an assistive device, used a hearing aid, used hearing protection).

OTHER OUTCOMES:
Mean value for hearing-specific health-related quality of life at eight weeks post baseline as measured by a series of study-specific questions, some of which are adapted from the Self Assessment of Communication | 8 weeks
  Participants rate the impact of hearing loss on various aspects of their lives, such as their emotional state and enjoyment of life.
Communication function with partner: Mean frequency and severity of communication-related challenges as measured by a series of study-specific questions at eight weeks post baseline | 8 weeks
  Frequency and difficulty of communication-related challenges resulting from hearing loss.
Mean confidence in communication management at eight weeks post baseline as measured by a series of study-specific questions | 8 weeks
  Participants rate their confidence in being able to manage their hearing loss and communication with family and other communication partners.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Marrone, PhD, Principal Investigator — University of Arizona
Locations (1):
- Mariposa Community Health Center, Nogales, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Marrone NL, Nieman CL, Coco L. Community-Based Participatory Research and Human-Centered Design Principles to Advance Hearing Health Equity. Ear Hear. 2022 Jul-Aug 01;43(Suppl 1):33S-44S. doi: 10.1097/AUD.0000000000001183. Epub 2020 Jun 13. PMID 35724253